CLINICAL TRIAL: NCT03974555
Title: Epidemiological Investigation and Cohort Study on Food Allergy in Children Aged 3 to 6 Years in Wenzhou and Taizhou Urban Areas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2018-06-214
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Food Hypersensitivity
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective

1. To investigate the status of food allergy among children aged 3 to 6 in Wenzhou and Taizhou urban areas.
2. To obtain the self-reported rate of parents or guardians of food allergy among children aged 3 to 6 in Wenzhou and Taizhou urban areas.
3. To obtain the prevalence of food allergy among children aged 3 to 6 in Wenzhou and Taizhou urban areas by conducting skin prick test (SPT), blood eosinophil (EOS) count, total immunoglobulin E (tIgE) measurement and serum specific IgE (sIgE) determination in children who self-reported food allergy, and conducting the open food challenge (OFC) if it is needed for further diagnosis.

Methods The preschool children aged 3 to 6 from kindergartens in Wenzhou and Taizhou urban areas were selected by cluster sampling and random sampling to conduct a preliminary screening questionnaire. Then telephone interviewe the children who had diseases or problems caused by certain food or certain types of food. Make them finish further food allergy questionnaires, SPT, EOS, tIgE detection, sIgE detection. SPT has 17 kinds of food allergens including milk, egg white, egg yolk, shrimp, crab, wheat, mackerel, perch, cod, peanut, cashew nut, soybean, peach, pineapple, mango, orange and kiwifruit. sIgE has 10 kinds of food allergens including milk, egg white, shrimp, crab, soybean, peanut, wheat, nut mixed group and food mixed group. Children whose results of SPT and/or sIgE didn't meet the diagnostic criteria and children whose results of SPT and sIgE were negative but its history strongly supported food allergy need to conduct OFC. Descriptive analysis and risk factor analysis were carried out on the results, and SPSS 18.0 statistical software was used in statistics analyzation.

ELIGIBILITY:
Inclusion Criteria:

* The date of birth is in the range of 2011.9.1-2015.8.31

Exclusion Criteria:

* The date of birth is not in the range of 2011.9.1-2015.8.31 or the children who's parents cannot cooperate

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preschool children aged 3 to 6 years in Lucheng District, Ouhai District of Wenzhou and Jiaojiang District and Huangyan District of Taizhou
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
the prevalence of food allergy | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Huan Dai, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Dai H, Wang F, Wang L, Wan J, Xiang Q, Zhang H, Zhao W, Zhang W. An epidemiological investigation of food allergy among children aged 3 to 6 in an urban area of Wenzhou, China. BMC Pediatr. 2020 May 14;20(1):220. doi: 10.1186/s12887-020-02115-8. PMID 32410652